CLINICAL TRIAL: NCT02848794
Title: Phase I/IIa, Single-Arm, Open Study of Apatinib and Irinotecan in Treating Patients With Recurrent High-grade Glioma
Brief Title: Apatinib and Irinotecan in Treating Patients With Recurrent High-grade Glioma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First People's Hospital of Lianyungang (Other)
Collaborators: Shandong Cancer Hospital and Institute (Other); The Affiliated Hospital of Qingdao University (Other); Yankuang Group General Hospital (Unknown); Lianyungang Hospital Affiliated Bengbu Medical College (Other); Suzhou Kowloon Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI-001
Record Dates: First submitted 2016-07-22; First posted 2016-07-28 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: High-grade Glioma
MeSH Terms: conditions — Glioma | interventions — apatinib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apatinib+Irinotecan (Experimental): Apatinib and irinotecan in treating patients with recurrent high-grade glioma,who have progressed on temozolomide, or radiotherapy alone, or combined with chemotherapy within 3 months after surgery .
  Interventions: Drug: Apatinib and Irinotecan

INTERVENTIONS:
Drug: Apatinib and Irinotecan — Patients were administered at apatinib (850mg po qd) and irinotecan(125mg/m2 d1,8) intravenously every three weeks for up to 6 cycles.Maintenance apatinib (500mg po qd) was administered until disease progression or unacceptable toxicity.

SUMMARY:
The study is aimed to evaluate the efficacy and safety of Apatinib and Irinotecan in patients with recurrent high-grade glioma.

DETAILED DESCRIPTION:
Gliomas account for almost 80% of primary malignant brain tumors, and glioblastoma is the most common subtype. Despite treatment with surgery, radiation, and chemotherapy(Temozolomide) almost all patients with glioma experience recurrence and the median survival for most patients is less than 2 years. In recurrent disease, salvage therapies have been limited and result in minimal improvement in OS. This overwhelming need for improved treatments has driven the development of novel drugs that target glioma biology, specifically anti-VEGF therapies.

Malignant gliomas are considered among the most angiogenic of cancers and are mostly fueled by vascular endothelial growth factor (VEGF) signaling via its endothelial tyrosine kinase receptor VEGF receptor 2 (VEGFR2). Levels of VEGF and its receptor are correlated with the histologic grade of gliomas, with the highest levels present in glioblastoma.Thus glioblastoma has emerged as an attractive tumor in which to conduct clinical trials of novel anti-VEGF agents, such as monoclonal antibodies and tyrosine kinase inhibitors.

Bevacizumab is a recombinant humanized monoclonal antibody that binds all VEGF isoforms, causing reduced tumor vascularization and inhibiting tumor growth. In a single-institute, phase II trial of patients with recurrent high-grade glioma, bevacizumab in combination with irinotecan demonstrated 46% 6-month PFS and 57% OR rates. Following on from the results of this study, another phase II trial was conducted to evaluate the safety and efficacy of bevacizumab alone and in combination with irinotecan, again showing promising results. On the basis this study, as well as a study by Kreisl and colleagues, FDA has approved to bevacizumab for patients with recurrent glioblastoma in 2009. Despite bevacizumab therapy, 6-month progression-free survival (PFS) for relapsed or progressive high-grade gliomas is 30.8% to 50.3%, and median overall survival (OS) is less than 42 week. Thus, recurrent high-grade gliomas remains a largely unmet medical need, which highlights the need for novel and effective therapies.

Apatinib is a small-molecule tyrosine kinase inhibitor (TKI) that highly selectively binds to and strongly inhibits vascular endothelial growth factor receptor 2 (VEGFR-2). Apatinib has been demonstrated as monotherapy prolongs OS in patients with gastric or gastroesophageal junction adenocarcinoma after two or more lines of chemotherapy with moderate, reversible, and easily managed adverse events.

The study is aimed to evaluate the efficacy and safety of Apatinib and Irinotecan in patients with recurrent high-grade glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-confirmed, high-grade glioma(WHO Ⅲ/Ⅳ) who have progressed on temozolomide, or radiotherapy alone, or combined with chemotherapy within 3 months after surgery .
2. With measurable or evaluable disease defined by RECIST 1.1 criteria by MRI scan.
3. Eastern Cooperative Oncology Group Performance Status (ECOG P.S.) of ≤ 2
4. Life expectancy ≥3 months.
5. No evidence of serious cardiopulmonary function damage, postoperative complication and hemorrhage on the baseline.
6. No history of cerebral embolism, cerebral hemorrhage and serious hypertension disease.
7. Recovery from the effects of prior therapy, including the following: 4 weeks from cytotoxic agents (except 6 weeks from nitrosoureas and mitomycin), radiotherapy and surgery.
8. Patients have adequate organ function as defined by the following criteria:

   * Hemoglobin (HGB) ≥90g/L
   * Absolute neutrophil count (ANC) ≥1.5×109/L
   * White blood cell (WBC) ≥3.0×109/L
   * Platelet count ≥80×109/L
   * Alanine aminotransferase(ALT) and Aspartate aminotransferase (AST) of ≤2.5 upper normal limitation (UNL) or ≤5 UNL in case of liver metastasis
   * Creatinine (Cr) of ≤1.25 UNL or creatinine clearance(Ccr) > 45 ml/min.
9. Patients will take contraceptive measures for the duration of the treatments and 8 weeks after the last treatment.
10. With written informed consent signed voluntarily by patients themselves.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Inadequately controlled hypertension (defined as systolic blood pressure > 140 and/or diastolic blood pressure > 90 mmHg on antihypertensive medications).
3. New York Heart Association (NYHA) Grade II or greater congestive heart failure.
4. Coronary heart disease greater than ClassⅠ;Ⅰ-level arrhythmia (including QT interval prolongation≥440 ms) together with ClassⅠcardiac dysfunction
5. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction).
6. Abnormal Coagulation (international normalized ratio>1.5, prothrombin time>UNL+4s,activated partial thromboplastin time>1.5 UNL), with tendency of bleeding.
7. Currently receive thrombolytic and anticoagulation therapy
8. History of pneumorrhagia(CTCAE grade ≥2 ) or other parts hemorrhage(CTCAE grade ≥3 ) within 4 weeks prior to treatment.
9. History of artery thrombosis and phlebothrombosis, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism, within 6 month prior to treatment.
10. Medical history of clinically significant thrombosis (bleeding or clotting disorder), excluding warfarin(1mg po qd) and aspirin(80-100mg po qd) for prevention under INR≤1.5.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to progression of disease. Estimated about 6 months
  The length of time from enrollment until the time of progression of disease (PFS, progression-free survival)

SECONDARY OUTCOMES:
Overall Survival (OS) | From enrollment to death of patients. Estimated about 1 year
  The length of time from enrollment until the time of death (OS, overall survival)
Objective Response Rate (ORR) | From enrollment to 2 months after treatment
  clinical response of treatment according to RESIST v1.1 criteria (ORR, objective response rate)
Disease Control Rate (DCR) | From enrollment to 2 months after treatment
  Disease control rate is defined as the number of patients with a best overall response of complete response (CR), partial response (PR), or stable disease (SD) based on RESIST v1.1 criteria.
Duration of Response（DOR） | From first documented CR or PR until disease progression or death(up to 1 year)
  As measured by RECIST 1.1 criteria and defined as the time from the first documented CR or PR until disease progression or death from any cause.
Quality of life (QOL) | up to 1 year
  Quality of life (QOL) will be measured using the EORTC QLQ-C30 questionnaires,which consists of 28 questions with answers that range from 1 (Not At All) to 4 (Very Much) and 2 questions that range from 1 (Very Poor) to 7 (Excellent)
Incidence of treatment-related adverse events | up to 1 year
  The incidence of treatment-related adverse events were graded with the use of the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First's People Hospital of Lianyungang, Lianyungang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang L, Liang L, Yang T, Qiao Y, Xia Y, Liu L, Li C, Lu P, Jiang X. A pilot clinical study of apatinib plus irinotecan in patients with recurrent high-grade glioma: Clinical Trial/Experimental Study. Medicine (Baltimore). 2017 Dec;96(49):e9053. doi: 10.1097/MD.0000000000009053. PMID 29245310